CLINICAL TRIAL: NCT02329834
Title: Open-label, Single-dose, Randomized, Two-way (Two-period) Crossover Study to Compare the Pharmacokinetics and Bioavailability of a Novel Furosemide Regimen Administered Subcutaneously Versus the Same Dose (80mg) Administered Intravenously in Subjects With Chronic Heart Failure
Brief Title: Crossover Study to Compare the Pharmacokinetics and Bioavailability of a Novel Furosemide Regimen Administered Subcutaneously vs. the Same Dose Administered Intravenously in Subjects With Chronic Heart Failure
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: scPharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: scP-01-002
Record Dates: First submitted 2014-12-22; First posted 2015-01-01 (Estimated); Results first posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Furosemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Sequence 1 (Experimental): Furosemide Injection Solution for subcutaneous administration (80mg) over 5 hours followed by i.v. Furosemide Injection, USP (80 mg)by i.v. bolus in second period
  Interventions: Drug: Fursemide Injection Solution for subcutaneous administration (80 mg); Drug: Furosemide Injection, USP
- Treatment Sequence 2 (Experimental): Furosemide Injection, USP (80 mg) by i.v. bolus, followed by Furosemide Injection Solution for subcutaneous administration (80mg) over 5 hours in second period.
  Interventions: Drug: Fursemide Injection Solution for subcutaneous administration (80 mg); Drug: Furosemide Injection, USP

INTERVENTIONS:
Drug: Fursemide Injection Solution for subcutaneous administration (80 mg) — Furosemide Injection Solution, 10mL of undiluted buffered furosemide solution (8mg/mL)
Drug: Furosemide Injection, USP — Furosemide Injection, USP (10mg/mL), 80 mg by intravenous administration.

SUMMARY:
The proposed study aims to compare the pharmacokinetics and bioavailability of intravenous and subcutaneous Furosemide. Although these regimens are not intended to be bioequivalent, they are both expected to achieve therapeutic plasma levels and induce effective diuresis.

The test formulation in this study is a buffered solution, Furosemide Injection Solution at 8 mg/mL at pH 7.4 (range 7.0 to 7.8) and is intended for SC injection according to the instructions in the protocol. A commercial formulation of Furosemide Injection, USP will serve as the reference drug in this study, which will be administered by IV bolus. It contains furosemide 10 mg/mL in solution at alkaline pH of 8.0 to 9.3 and is marketed for IV and IM injection.

The objectives of this study are:

* To characterize the pharmacokinetics of furosemide administered by continuous subcutaneous infusion using a biphasic delivery profile.
* To estimate the absolute bioavailability of furosemide administered by continuous subcutaneous infusion compared with an equivalent dose of furosemide administered by intravenous bolus administration.

DETAILED DESCRIPTION:
This study will be an open-label, single-center, single-dose, randomized, two-way (two-period) crossover study in 16 adult subjects previously diagnosed with mild to moderate heart failure (NYHA class II/III) being treated concomitantly with oral furosemide therapy at a dose of ≥ 40 mg/day. Each subject will complete Screening, Baseline, Treatment, and Follow-Up Phases. The Screening Phase will be conducted on an outpatient basis between 14 and 3 days prior to Baseline. Subjects will be instructed to maintain a < 2 gm sodium diet within 3 days prior to Baseline. Baseline (Day 0) consists of clinical research unit (CRU) admission and final qualification assessments. The Treatment Phase will comprise two crossover periods separated by a 7-day outpatient fluid re-equilibration washout. Following CRU admission, subjects will discontinue oral furosemide at least 24 hours prior to administration of study drug for each Crossover Period. Subjects will be randomly assigned in a 1:1 ratio to 1 of 2 treatment sequences to receive both intravenous (IV) and subcutaneous (SC) furosemide in Crossover Periods (i.e., IV followed by SC or vice versa). Subjects will remain domiciled in the CRU for each Crossover Period during the Treatment Phase through 24 hours after administration of study drug, after which time they will be discharged if safety parameters are acceptable to the Investigator. Oral furosemide therapy will be re-initiated at discharge after Crossover Period 1 (i.e., during the 7-day fluid re-equilibration washout) and after Crossover Period 2. The Follow-Up Phase will occur 7 days (± 1) after discharge from the CRU following Crossover Period 2, completing subjects' study participation.

ELIGIBILITY:
Inclusion Criteria:

* An Institutional Review Board (IRB) approved informed consent is signed and dated prior to any study-related activities.
* Male and female subjects ≥18 years of age, with body volume and weight <130 kg and body mass index (BMI) <38 kg/m2
* Females will be non-pregnant, non-lactating, and post-menopausal, surgically sterile (e.g., tubal ligation, hysterectomy), or use TWO (2) of the following forms of contraception: IUD, IUD with spermicide, female condom with spermicide, contraceptive sponge with spermicide, an intravaginal system, diaphragm with spermicide, cervical cap with spermicide, a male sexual partner who agrees to use a male condom with spermicide, a sterile sexual partner, OR abstinence
* History of at least 3 months treated heart failure (NYHA class II/III) with presence of symptoms of chronic volume overload requiring ongoing treatment with oral furosemide at a dose of ≥ 40 mg per day for at least 30 days prior to baseline
* NT-proBNP > 300 pg/mL or BNP > 100 pg/mL
* Agrees to abstain from using alcohol, caffeine-containing products, and tobacco-/nicotine-containing products through CRU discharge (period 2).
* Able to participate in the study in the opinion of the investigator
* Has the ability to understand the requirements of the study and is willing to comply with all study procedures

Exclusion Criteria:

* Acute Decompensated Heart Failure (ADHF) or recent history of hospitalization for heart failure in the last 4 weeks
* Worsening of signs or symptoms of heart failure in the two weeks prior to the Screening, or those expected to require intravenous loop diuretics or in-patient treatment for heart failure during the study
* Systolic BP (SBP) < 90 mm Hg
* Temperature > 38°C (oral or equivalent) or sepsis or active infection requiring IV anti-microbial treatment
* Serum sodium < 130 mEq/L and Serum potassium < 3.0 mEq/L
* Significant other cardiac abnormalities which may interfere with study participation or study assessments
* Current or planned treatment during the study with any IV therapies, including inotropic agents, vasopressors, levosimendan, nesiritide or analogues; or mechanical support (intra-aortic balloon pump, endotracheal intubation, mechanical ventilation, or any ventricular assist device)
* Diagnosed with Type I diabetes mellitus or Type II diabetes requiring insulin therapy
* Presence or need for urinary catheterization, urinary tract abnormality, or disorder interfering with urination
* Impaired renal function, defined as an estimated glomerular filtration rate (eGFR) on admission < 45 mL/min/1.73m2, calculated using the simplified Modification of Diet in Renal Disease (sMDRD) equation
* Indication of moderate-to-severe hepatic dysfunctions as determined by the investigator
* Administration of intravenous radiographic contrast agent within 72 hours prior to Screening or acute contrast-induced nephropathy at the time of Screening
* Major surgery within 30 days prior to Screening
* Administration of an investigational drug or implantation of investigational device, or participation in another interventional trial, within 30 days prior to Screening
* Any surgical or medical condition which in the opinion of the investigator may interfere with participation in the study or which may affect the outcome of the study
* Positive test for hepatitis B, hepatitis C, or HIV at Screening
* Positive urine drug screen at Screening or Baseline
* Concomitant use of any drugs known to interact with furosemide
* History of alcohol abuse within 6 months prior to screening, as determined by the Investigator
* Positive alcohol breath test on admission to the CRU
* History of severe allergic or hypersensitivity reactions to furosemide
* Donation of greater than 100 mL of either whole blood or plasma within 30 days prior to study drug administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-04; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce G. Rankin, DO, CPI, MRO, FACOFP, Principal Investigator — Avail Clnical Research, LLC
Locations (1):
- Avail Clinical Research, LLC, DeLand, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 6 subjects did not meet inclusion/exclusion criteria after signing informed consent.
  * 2 subjects did not meet the inclusion criteria of BNP>100pg/ml
  * 2 subjects met the exclusion criterion: Impaired renal function, defined as an eGFR on admission <45 mL/min/1.73m2
  * 1 subject withdrew consent
  * 1 subject was excluded by the investigator due to High Creatine Kinase
Groups:
- Treatment Sequence 1 (SC Period 1; IV Period 2): Furosemide Injection Solution for subcutaneous administration (80mg) over 5 hours followed by i.v. Furosemide Injection, USP (80 mg)by i.v. bolus in second period
  Fursemide Injection Solution for subcutaneous administration (80 mg): Furosemide Injection Solution, 10mL of undiluted buffered furosemide solution (8mg/mL)
  Furosemide Injection, USP: Furosemide Injection, USP (10mg/mL), 80 mg by intravenous administration.
- Treatment Sequence 2 (IV Period 1; SC Period 2): Furosemide Injection, USP (80 mg) by i.v. bolus, followed by Furosemide Injection Solution for subcutaneous administration (80mg) over 5 hours in second period.
  Fursemide Injection Solution for subcutaneous administration (80 mg): Furosemide Injection Solution, 10mL of undiluted buffered furosemide solution (8mg/mL)
  Furosemide Injection, USP: Furosemide Injection, USP (10mg/mL), 80 mg by intravenous administration.
Period: Overall Study
Arm/Group | Treatment Sequence 1 (SC Period 1; IV Period 2) | Treatment Sequence 2 (IV Period 1; SC Period 2)
Started | 8 | 9
Completed | 7 | 9
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT): All randomized subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Sequence 1 (SC Period 1; IV Period 2) | Treatment Sequence 2 (IV Period 1; SC Period 2) | Total
Number analyzed (Participants) | 8 | 9 | 17
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72.4 (7.3) | 64.1 (9.4) | 68 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 6 | 9 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 8 | 7 | 15
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 9 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
NYHA Class [Count of Participants; unit: Participants] — New York Heart Association Classification
  * Class I: No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea.
  * Class II: Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea.
  * Class III: Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or dyspnea.
  * Class IV: Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest that worsen with physical activity.
  Participants
    NYHA II | 7 | 6 | 13
    NYHA III | 1 | 3 | 4
Participants with History of Ischemic Heart Disease [Count of Participants; unit: Participants]
  Ischemic | 2 | 4 | 6
  Non-Ischemic | 6 | 5 | 11
Participants with History of Hypertension [Count of Participants; unit: Participants] | 8 | 9 | 17
Participants with History of Arrhythmia [Count of Participants; unit: Participants] | 6 | 8 | 14
Participants with History of Acute Myocardial Infarction [Count of Participants; unit: Participants] | 4 | 8 | 12
BMI [Mean (Standard Deviation); unit: kg/m^2] | 31.5 (4.6) | 30.9 (4.8) | 31 (4.6)
BMI [Count of Participants; unit: Participants]
  <=30kg/m^2 | 2 | 3 | 5
  >30kg/m^2 | 6 | 6 | 12
proBNP [Mean (Standard Deviation); unit: pg/mL] | 891 (805) | 903.2 (1037.5) | 897 (906.5)
Participants with History of Diabetes [Count of Participants; unit: Participants] | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Cmax
Description: Maximum observed plasma concentration of Furosemide
Time Frame: 0, 5 min, 15 min, 30 min, 45 min, 60 min, 1.5 hours, 2 hours, 2:05 min, 2:15 min, 2:30 min, 2:45 min, 3 hours, 3:30 min, 4, 5, 6, 8, 10, 12, 14, and 16 hours post-dose
Population: PK Population: All randomized subjects who receive study drug and have sufficient samples collected for estimation of pharmacokinetic parameters
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- IV Furosemide: Pharmacokinetic Assessments after a successful IV dosing regimen
- SC Furosemide: Pharmacokinetic Assessments after a successful SC dosing regimen
Arm/Group | IV Furosemide | SC Furosemide
Number analyzed (Participants) | 15 | 15
ng/mL | 8580 (2540) | 2040 (449)

2. Primary Outcome: Tmax
Description: Time to achieve maximum observed Furosemide plasma concentration
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | IV Furosemide | SC Furosemide
Number analyzed (Participants) | 15 | 15
hours | 2.08 [0.08 to 2.08] | 4 [1 to 5.08]

3. Primary Outcome: AUClast
Description: The area under the plasma concentration versus time curve from time 0 (pre-dose) to the last quantifiable time point.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | IV Furosemide | SC Furosemide
Number analyzed (Participants) | 15 | 15
h*ng/mL | 13000 (4050) | 13000 (4000)
Statistical Analysis 1: Comparison: IV Furosemide; Test type: Equivalence — 90% Confidence Interval 80<ratio of AUC<125. The FDA guided Bioequivalence limit of 80 to 125% for the ratio of the product averages has been adopted for use of an average BE criterion; % diff Geometric Least Squared Mean = 99.50, 90% CI 2-sided [94.77 to 104.75]

4. Primary Outcome: AUCinf
Description: The area under the plasma concentration-time curve from time 0 (pre-dose) to time of last measurable plasma concentration.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | IV Furosemide | SC Furosemide
Number analyzed (Participants) | 15 | 15
h*ng/mL | 13200 (4170) | 13100 (4010)
Statistical Analysis 1: Comparison: IV Furosemide; Test type: Other; % Diff Geometric Least Squared Mean = 99.65, 90% CI 2-sided [94.79 to 104.75]

5. Primary Outcome: AUCext
Description: The percentage of AUC that is extrapolated beyond the last measurable concentration
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of AUC
Arm/Group | IV Furosemide | SC Furosemide
Number analyzed (Participants) | 15 | 15
percentage of AUC | 0.912 (0.631) | 1.05 (1.29)

6. Primary Outcome: λz
Description: Apparent plasma terminal-phase elimination rate constant
Time Frame: 24 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 1/h
Arm/Group | IV Furosemide | SC Furosemide
Number analyzed (Participants) | 15 | 15
1/h | 0.277 (0.0365) | 0.238 (0.0732)

7. Primary Outcome: t 1/2
Description: Terminal-phase half life
Time Frame: 24 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | IV Furosemide | SC Furosemide
Number analyzed (Participants) | 15 | 15
hours | 2.55 (0.339) | 3.16 (0.911)

8. Primary Outcome: Volume of Distribution, Terminal Phase
Description: Systemic Volume of distribution, terminal phase for IV furosemide and Apparent Volume of distribution, terminal phase for SC furosemide
Time Frame: 24 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Litres
Arm/Group | IV Furosemide | SC Furosemide
Number analyzed (Participants) | 15 | 15
Litres | 24.4 (9.15) | 28.5 (5.28)

9. Primary Outcome: CL
Description: Systemic Clearance for IV furosemide and Apparent Systemic Clearance for SC furosemide
Time Frame: 24 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: liter per hour
Arm/Group | IV Furosemide | SC Furosemide
Number analyzed (Participants) | 15 | 15
liter per hour | 6.71 (2.31) | 6.71 (2.21)

ADVERSE EVENTS:
Time Frame: Day 0 through Day-19 visit
Description: An AE is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.
  An SAE is any AE occurring at any dose that results in any of the following outcomes:
  * Death
  * Life threatening AE
  * Inpatient hospitalization or prolongation
  * Disability
  * Congenital anomaly or birth defect
  * Any important medical events based on investigator's clinical judgement.
Groups:
- During Washout or Follow-up: During washout or follow-up periods
Arm/Group | IV Furosemide | SC Furosemide | During Washout or Follow-up
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 2/16 | 10/16 | 5/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IV Furosemide (N=16) | SC Furosemide (N=16) | During Washout or Follow-up (N=16)
Application site erythema (General disorders) | 1 | 8 | 0
Application site edema (General disorders) | 0 | 7 | 0
Nodule (General disorders) | 0 | 0 | 1
BNP elevated (Investigations) | 0 | 0 | 1
Peripheral pulse decreased (Investigations) | 0 | 0 | 1
Total CK elevated (Investigations) | 0 | 0 | 1
Troponin elevated (Investigations) | 0 | 0 | 1
COPD (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No